CLINICAL TRIAL: NCT07223814
Title: Bleximenib or Placebo in Combination With Standard Induction and Consolidation Therapy Followed by Maintenance for the Treatment of Patients With Newly Diagnosed KMT2A-rearranged or NPM1-mutant Acute Myeloid Leukemia Eligible for Intensive Chemotherapy: a Double-blind Phase 3 Study
Brief Title: Bleximenib in Combination With Standard Induction and Consolidation Therapy Followed by Maintenance for Treatment of Patients With Acute Myeloid Leukemia (AML)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: German-Austrian Acute Myeloid Leukemia Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOVON 181 AML; 2025-522767-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; adult; newly diagnosed AML; NPM1; KMT2A
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; Idarubicin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Standard of care treatment plus bleximenib and also maintenance treatment with bleximenib (Experimental): Bleximenib in combination with remission induction and consolidation therapy, followed by bleximenib maintenance therapy. Treatment will continue until PD, unacceptable toxicity or other protocol defined criteria for discontinuation (whichever comes first)
  Interventions: Drug: Bleximenib; Drug: Cytarabine; Drug: Daunorubicin or Idarubicin
- Arm 2: Standard of care treatment plus bleximenib and maintenance treatment with a placebo. (Experimental): Bleximenib in combination with remission induction and consolidation therapy, followed by placebo maintenance therapy. Treatment will continue until PD, unacceptable toxicity or other protocol defined criteria for discontinuation (whichever comes first)
  Interventions: Drug: Bleximenib; Drug: Cytarabine; Drug: Daunorubicin or Idarubicin; Drug: Placebo
- Arm 3: Standard of care treatment plus a placebo and maintenance treatment with a placebo. (Placebo Comparator): Placebo comparator in combination with remission induction and consolidation therapy, followed by placebo maintenance therapy . Treatment will continue until PD, unacceptable toxicity or other protocol defined criteria for discontinuation (whichever comes first)
  Interventions: Drug: Cytarabine; Drug: Daunorubicin or Idarubicin; Drug: Placebo

INTERVENTIONS:
Drug: Bleximenib — Participants will receive bleximenib
  Arms: Arm 1: Standard of care treatment plus bleximenib and also maintenance treatment with bleximenib; Arm 2: Standard of care treatment plus bleximenib and maintenance treatment with a placebo.
Drug: Cytarabine — Participants will receive Cytarabine
Drug: Daunorubicin or Idarubicin — Participants will receive Daunorubicin or Idarubicin
Drug: Placebo — Participants will receive Placebo
  Arms: Arm 2: Standard of care treatment plus bleximenib and maintenance treatment with a placebo.; Arm 3: Standard of care treatment plus a placebo and maintenance treatment with a placebo.

SUMMARY:
The current standard of care treatment for adult patients with acute myeloid leukemia (AML) consists of chemotherapy and, if indicated, donor stem cell transplantation.

Bleximenib blocks the interaction between a protein called menin and another protein called KMT2A in the leukemia cells. When this interaction is disrupted in AML with mutations in the NPM1 or KMT2A gene, bleximenib can cause leukemia cells to die.

The main objective is to assess if treatment with bleximenib, when added to chemotherapy treatment will improve treatment outcome in adult participants with newly diagnosed AML who present with mutations in the NPM1 or KMT2A genes.

This is a randomized, double-blind, placebo-controlled, phase 3 clinical trial. All of the participants will receive standard chemotherapy treatment, combined with either bleximenib or a placebo. A placebo is a substance that looks like the study medicine but has no active ingredients (e.g., a sugar pill). In a double blind trial neither the participant nor the doctor know if placebo or active study drug is given.

After the end of the protocol treatment there will be an observational follow-up of 4 years from the time of inclusion of the last patient. The results of the different treatment groups will be compared.

875 previously untreated patients with AML with a specific change in the DNA of the leukemia cells (a KMT2A rearrangement or a NPM1 mutation) will be included. Participants must be 18 years or older and considered eligible for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age (or the legal age of majority in the jurisdiction in which the study is taking place, whichever is greater) at the time of informed consent.
2. New diagnosis of AML (≥10% blasts in BM or peripheral blood) with mutated NPM1 or with recurring rearrangements involving KMT2A according to ICC 2022 criteria.
3. Considered eligible for intensive chemotherapy.
4. WHO/ECOG performance status ≤2.
5. Adequate renal and hepatic functions prior to randomization.

Exclusion Criteria:

1. Prior (chemo-)therapy for AML, including prior treatment with hypomethylating agents
2. Known active leukemic involvement of the central nervous system (CNS).
3. Recipient of solid organ transplant.
4. Cardiac disease:

   1. Any of the following within 6 months of randomization: myocardial infarction, uncontrolled/unstable angina, congestive heart failure (NYHA Class III or IV), uncontrolled or symptomatic arrhythmias, stroke, or transient ischemic attack.
   2. QTc interval using Fridericia's formula (QTcF) ≥470 ms. Prolonged QTc interval associated with bundle branch block or pacemaking is permitted.
   3. Left ventricular ejection fraction (LVEF) <40% by ECHO or MUGA scan obtained within 28 days prior to the start of study treatment.
   4. Previously received cumulative dose of any combination of anthracyclines or anthracenediones of ≥500 mg/m2.
5. Chronic respiratory disease requiring supplemental oxygen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 875 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) in adult patients with newly diagnosed NPM1m or KMT2Ar AML eligible for intensive chemotherapy | Up to 4 years and 5 months
  To assess if treatment with bleximenib, as compared with placebo, in combination with remission induction chemotherapy, prolongs event-free survival (EFS) measured from the time from randomization to failure to achieve CR after remission induction, hematologic relapse after achieving CR, or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) in adult patients with newly diagnosed NPM1m or KMT2Ar AML eligible for intensive chemotherapy | Up to 7 years and 10 months
  To assess if treatment with bleximenib, as compared with placebo, in combination with remission induction and consolidation chemotherapy, followed by maintenance therapy, prolongs overall survival (OS) measured from randomization to death due to any cause.
Rates of CR, CRh, CRi in adult patients with newly diagnosed NPM1m or KMT2Ar AML eligible for intensive chemotherapy | Up to 7 years and 10 months
  Defined as the proportion of participants achieving a given response after induction cycle 1 and after induction cycle 2.
Prolongation of CR (DoCR) in adult patients with newly diagnosed NPM1m or KMT2Ar AML eligible for intensive chemotherapy | Up to 4 years and 5 months
  Defined as the time from achieving first response of CR to hematologic relapse or death from any cause, whichever occurs first.
Percentage of participants undergoing an allo-SCT in adult patients with newly diagnosed NPM1m or KMT2Ar AML eligible for intensive chemotherapy | Up to 7 years and 10 months
  To assess the percentage of participants undergoing an allo-SCT as part of protocol treatment

IPD SHARING:
Plan to Share IPD: Yes
According to the current publication policy the protocol and Statistica! Analysis Plan ( SAP) will be shared. The principal lnvestigators can be contacted for IPD sharing after the publication of the study results. According to 'HOVON sample and/or Data request Form' theHOVON director; chair of theHOVON Acute Myeloid Leukemie working group, the study PI and Coordinating lnvestigator should approve data/sample sharing.
Supporting Information: Study Protocol, SAP
Time Frame: After the publication of primary endpoint analysis